CLINICAL TRIAL: NCT00993018
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-42160443 in Subjects With Diabetic Painful Neuropathy, Followed by a Double-Blind Safety Extension and an Open-Label Safety Extension
Brief Title: A Study of Effectiveness and Safety of JNJ-42160443 in Patients With Diabetic Painful Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistic reasons associated with the FDA-imposed clinical hold.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR016438; 42160443NPP2002 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); 2008-007676-13 (EudraCT Number)
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetic Neuropathy; Diabetic painful neuropathy; JNJ-42160443; Neuropathic pain; Pain; Pharmacokinetics
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia; Pain | interventions — fulranumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- JNJ-42160443 (1 mg) (Experimental): JNJ-42160443 1 mg will be administered as a single, subcutaneous injection every 28 days for up to first 52 weeks in the blinded fashion and then every 28 days for up to an additional 52 weeks in the open-label fashion.
  Interventions: Drug: JNJ-42160443 (1 mg)
- JNJ-42160443 (3 mg) (Experimental): JNJ-42160443 3 mg will be administered as a single, subcutaneous injection every 28 days for up to first 52 weeks in the blinded fashion and then every 28 days for up to an additional 52 weeks in the open-label fashion.
  Interventions: Drug: JNJ-42160443 (3 mg)
- JNJ-42160443 (10 mg) (Experimental): JNJ-42160443 10 mg will be administered as a single, subcutaneous injection every 28 days for up to first 52 weeks in the blinded fashion and then every 28 days for up to an additional 52 weeks in the open-label fashion.
  Interventions: Drug: JNJ-42160443 (10 mg)
- Placebo (Placebo Comparator): Placebo will be administered as a single, subcutaneous injection every 28 days for up to 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42160443 (1 mg) — JNJ-42160443 1 mg will be administered as a single, subcutaneous injection every 28 days for up to first 52 weeks in the blinded fashion and then every 28 days for up to an additional 52 weeks in the open-label fashion.
  Arms: JNJ-42160443 (1 mg)
Drug: JNJ-42160443 (3 mg) — JNJ-42160443 3 mg will be administered as a single, subcutaneous injection every 28 days for up to first 52 weeks in the blinded fashion and then every 28 days for up to an additional 52 weeks in the open-label fashion.
  Arms: JNJ-42160443 (3 mg)
Drug: JNJ-42160443 (10 mg) — JNJ-42160443 10 mg will be administered as a single, subcutaneous injection every 28 days for up to first 52 weeks in the blinded fashion and then every 28 days for up to an additional 52 weeks in the open-label fashion.
  Arms: JNJ-42160443 (10 mg)
Drug: Placebo — Patients will receive single injection of matching placebo every 28 days for up to 52 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy, safety and tolerability of multiple doses of JNJ-42160443 when administered as a single, subcutaneous injection every 28 days to patients with diabetic painful neuropathy (a disease condition in diabetic patients that affects all peripheral nerves including pain fibers, motor neurons and the autonomic nervous system).

DETAILED DESCRIPTION:
This is a multicenter (study conducted at multiple sites), randomized (the study medication is assigned by chance), double-blind (neither investigator nor the patient knows the treatment that the patient receives), placebo-controlled (an inactive substance that is compared with the study medication to test whether the study medication has a real effect in clinical study), dose-ranging study (study carried out at different doses) to evaluate the analgesic efficacy, safety, and tolerability of multiple doses of JNJ-42160443 in patients with neuropathic pain, followed by a double-blind safety extension and an open-label (all people know the identity of the intervention) safety extension. The study will consist of 5 sequential phases: 1) screening, 2) a 12-week double-blind efficacy, 3) a 40-week double-blind safety extension, 4) a 52-week open-label safety extension, and 5) a 26-week post-treatment/follow-up. After the screening phase, patient randomization will be stratified by current pain medication use (patients who are currently using or who are not currently using permitted pain medication). The planned doses for the double-blind efficacy phase and double blind safety extension phase are placebo, JNJ-42160443 1, 3, or 10 mg administered as a single, subcutaneous injection every 28 days. Safety assessment will include adverse events, injection site evaluations, clinical laboratory tests, electrocardiogram, vital signs, physical examinations, neurological examinations, and joint safety which will be monitored throughout the study. The total study duration (including all the 5 phases) will be approximately 131 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neuropathic pain (pain persistent for greater than 6 months) that is moderate to severe in the opinion of the investigator
* Currently taking neuropathic pain medication limited to maximal allowed doses according to guidelines provided, but are not adequately controlled by standard of care
* Currently not taking neuropathic pain medications because they are intolerable to, or not willing to use, standard of care
* Mean average pain intensity score of at least 5, but less than 10, over 7 consecutive days on an 11-point numerical rating scale
* Pain due to bilateral peripheral neuropathy caused by type 1 or type 2 diabetes mellitus
* Required to have stable glycemic control

Exclusion Criteria:

* Patients with severe diabetic neuropathy defined by severe autonomic dysfunction or blood pressure instability Separate pain condition (e.g., joint osteoarthritis) that is more severe than their pain due to their diagnosis of Diabetic Peripheral Neuropathy
* Patients with evidence of another neuropathic pain not under the study, such as pain resulting from post-traumatic neuralgia, post-surgical neuropathy, complex regional pain, sensory neuropathies or pain caused by radiation, chemotherapy, alcohol, Human Immunodeficiency Virus (HIV) infection
* Major surgeries, trauma, and non-healing wounds/ulcers within 3 months prior to study medication
* History of severe traumatic brain injury within the past 15 years
* Other peripheral neuropathy, parasthesia or dyesthesia or previously diagnosed neurological condition causing these symptoms not related with diabetic painful neuropathy under study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Average pain intensity | Baseline to Week 13
  The mean of the daily evening assessment of average pain intensity is measured by using 11-point numerical rating scale (NRS), where 0 = no pain and 10 = pain as bad as the patient can imagine.

SECONDARY OUTCOMES:
Pain at its worst | Baseline to Week 13
  The assessment of pain at its worst in the past 24 hours will be performed once daily, in the evening, using an 11-point numerical rating scale (NRS), where 0 = no pain and 10 = pain as bad as the patient can imagine.
Brief Pain Inventory | Up to Week 105
  The Brief Pain Inventory short form (BPI-SF) includes 4 items assessing pain intensity (pain intensity subscales) and 7 items assessing how much pain has interfered with daily activities (pain interference subscales). The intensity of pain is assessed with 4 items using an 11-point NRS from 0 = no pain to 10 = higher severity of pain. This assessment will be conducted on daily basis.
Neuropathic pain symptom inventory (NPSI) | Up to Week 105
  The NPSI contains 12 questions designed to evaluate the different symptoms of neuropathic pain. The questions make up the following 5 subscales: burning (superficial) spontaneous pain, pressing (deep) spontaneous pain, paroxysmal pain, evoked pain and paresthesia/dysesthesia. Subscale scores can be derived from averaging the scores from the item scores that make up the subscales, ranging from 0 to 10. A total intensity score is the sum of the subscale scores, ranging from 0 to 100. Higher scores indicate worse pain. This assessment will be conducted on daily basis.
Patient Global Impression of Change (PGIC) | Up to week 105
  The patient will be asked to rate their change in their neuropathic pain with the following responses: very much improved, much improved, minimally improved, not changed, minimally worse, much worse, or very much worse. This assessment will be conducted on daily basis.
Number of patients with adverse events | Up to week 105 and 26 weeks after the last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L. L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (23):
- United States (23):
  - Jonesboro, Arkansas
  - Fresno, California
  - La Jolla, California
  - Long Beach, California
  - Redondo Beach, California
  - Tustin, California
  - Walnut Creek, California
  - Bradenton, Florida
  - Palm Beach Gardens, Florida
  - Baltimore, Maryland
  - Albany, New York
  - Syracuse, New York
  - Winston-Salem, North Carolina
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Greer, South Carolina
  - Tullahoma, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Renton, Washington